CLINICAL TRIAL: NCT03778840
Title: Prospective Study of Incidence and Risk Factors of Infections and of Replacement Therapy With Intravenous Immunoglobulins for Secondary Immunodeficiency in Patients With Autoimmune Diseases Treated With Rituximab
Brief Title: Study of Infections in Patients With Autoimmune Diseases Treated With Rituximab
Acronym: EXPRIME
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Grifols Biologicals, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018_06; 2018-A00188-47 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-09-18; First posted 2018-12-19 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Autoimmune Diseases
Keywords: Infections; immunoglobulins; secondary immunodeficiency; rituximab
MeSH Terms: conditions — Autoimmune Diseases; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rituximab is a very effective drug used to treat many inflammatory diseases. These diseases include, for example, rheumatoid arthritis, multiple sclerosis and systemic autoimmune diseases.

The major drawback of this drug is the risk of infection, which are favored by the direct effect of rituximab on the immune system. The risk of infection is one of the major reason not to prescribe or withdraw rituximab in several patients. However, many questions remain unanswered regarding the proportion and risk factors of infection or immunodeficiency induced by rituximab. Better understanding of these issues will help prescribing rituximab and properly monitor patients during their treatment. Moreover, as treatment with substitutive immunoglobulins might be a solution to decrease the risk of infections in those patients, it is very important to better characterize the risk and risk factors of rituximab-associated infection. The present study aims to answer these questions.

ELIGIBILITY:
Inclusion Criteria:

* Patient initiating treatment with RTX, delivered by the central pharmacy of Lille University Hospital
* Inpatient or outpatient at Lille University Hospital (in one of the following departments: internal medicine, rheumatology, neurology, dermatology, pneumology) and monitored every three months as part of routine care (as part of the surveillance of induction of RTX treatment)
* Patient with one of the following autoimmune diseases, defined by international criteria

Exclusion Criteria:

* Treatment with rituximab for a malignancy or a transplant reject
* Pregnant or lactating women
* People in emergency
* Administrative reasons: inability to receive informed information, inability to participate in the entire study, lack of coverage by the social security system, refusal to sign consent
* Persons deprived of their liberty
* People unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients included in the study will be the patients beginning a cure of RTX prescribed within the framework of the treatment of their inflammatory disease or dysimmunitaire chronic.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of a serious infection event [SIE] in patient with an autoimmune disease treated with rituximab | Within 12 months after inclusion
  A serious infection event [SIE] defined as any infection which led to hospitalization and/or death and/or required treatment with intravenous antibiotic/antiviral drugs

SECONDARY OUTCOMES:
Hypogammaglobulinemia | Within 12 months after inclusion
  defined by immunoglobulin (Ig) G <6g / L.
Replacement therapy with immunoglobulins | Within 12 months after inclusion
  Start of an immunoglobulins therapy to replace gammaglobulins
Hypersensitivity skin reaction secondary to RTX injection. | Within 12 months after inclusion
  Attack rate of cutaneous hypersensitivity reactions after RTX injection in patients with dysimmune disease.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent SOBANSKI, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Claude Huriez, CHU, Lille, France